CLINICAL TRIAL: NCT04977674
Title: Investigating Glutamate and Opioid Mechanisms of Antidepressant Response to Ketamine
Brief Title: Glutamate and Opioid Mechanisms of Antidepressant Response to Ketamine
Acronym: GO-MARK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MR/T028084/1
Record Dates: First submitted 2021-07-01; First posted 2021-07-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: ketamine; naltrexone; glutamate; opioid; major depressive disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Naltrexone; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Visit 1) Naltrexone + Ketamine, Visit 2) Placebo + Ketamine (Experimental): Participants randomly assigned to arm A:
  VISIT 1) Naltrexone 50mg before the administration of ketamine 0.5mg/kg.
  VISIT 2) Placebo before the administration of ketamine 0.5mg/kg.
  Study visits are separated by 14-28 days.
  Interventions: Drug: Naltrexone; Drug: Placebo; Drug: Ketamine
- B: Visit 1) Placebo + Ketamine, Visit 2) Naltrexone + Ketamine (Experimental): Participants randomly assigned to arm B:
  VISIT 1) Placebo before the administration of ketamine 0.5mg/kg.
  VISIT 2) Naltrexone 50mg before the administration of ketamine 0.5mg/kg.
  Study visits are separated by 14-28 days.
  Interventions: Drug: Naltrexone; Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: Naltrexone — Pre-treatment with naltrexone 45 min before the ketamine infusion.
Drug: Placebo — Pre-treatment with placebo 45 min before the ketamine infusion.
Drug: Ketamine — Participants receive intravenous ketamine infusion (0.5 mg/kg over 40 min) at both study visits.

SUMMARY:
The overarching aim of this research is to determine the acute effects of ketamine on brain glutamate, functional connectivity and cerebral blood flow in treatment-resistant depression, explore whether the effects are attenuated by the opioid receptor antagonist naltrexone and relate these findings to antidepressant response.

DETAILED DESCRIPTION:
The study is a randomised, double-blind, crossover design with two treatment conditions: oral placebo or oral naltrexone preceding ketamine infusion during neuroimaging in subjects with treatment-resistant depression.

Each subject will participate in two imaging sessions on two separate days. Each subject will receive a dose of ketamine (IV infusion, 0.5 mg/kg over 40 minutes) during each scan. Subjects will receive either oral placebo or naltrexone 50 mg, 45 minutes before the initiation of each of the ketamine infusions.

ELIGIBILITY:
The following inclusion criteria will apply:

* Right-handed participants between the ages of 18 and 50 years inclusive.
* Able to provide informed written consent
* Fulfil Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5) criteria for a primary diagnosis of current single or recurrent episodes of MDD of at least moderate severity but without psychotic features as defined on the MINI 7.0. Positive and primary diagnoses on the MINI 7.0 will be subject to confirmation at clinical interview by a psychiatrist.
* 17-item HAM-D score ≥ 18.
* Have failed to respond to 2 or more antidepressants prescribed at minimum effective dose for at least 6 weeks OR at least 1 antidepressant prescribed at the minimum effective dose for at least 6 weeks AND a course of evidence-based psychotherapy given for at least 6 sessions.
* The subject is off all drugs likely to interact with glutamate or opioid system at least 14 days before starting the study (antipsychotics, anticonvulsants, mood stabilisers, gabapentinoids, opiates, opioid agonists/antagonists/combinations and stimulants). There are two exceptions. The first is any regular antidepressant(s) the subject may be taking (apart from MAOIs that are not permitted). Second, is short acting benzodiazepines or hypnotics for distressing anxiety or insomnia (up to 72 hours prior to each MRI scan).
* The subject has a resting pulse ≥51 bpm and ≤100 bpm at the screening visit. For subjects in good physical condition, the lower limit is ≥45 bpm.
* The subject has a resting systolic blood pressure ≥91 mmHg and ≤140 mmHg and a resting diastolic blood pressure ≥51 mmHg and ≤90 mmHg at the screening visit. An out-of-range resting systolic blood pressure may be repeated once if a medically valid reason is present, for example, the subject suffers from white-coat hypertension or has just come from low outdoor temperatures or experienced stress (e.g. late arrival). The medically valid reason must be documented and signed by the investigator.
* Body Mass Index (BMI) of 18 to 30 kg/m2 inclusive and a total body weight 50-100 kg at the screening visit.
* Able to attend interviews and tolerate MRI scanning procedures.

The following exclusion criteria will apply:

* Diagnosis of bipolar disorder or psychotic disorder on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
* A first-degree relative with bipolar disorder, schizoaffective disorder, or schizophrenia, with the potential participant younger than 33 years (ie, still at age of risk for a psychotic disorder).
* Personal history of a ≥ 1 suicide attempt in the past year, or active ideation with plan and intent defined using the C- SSRS ("Suicidal Behaviour" section and question 5) alongside confirmation at clinical interview with a psychiatrist.
* Diagnosis of drug or alcohol dependence syndrome (defined as meeting DSM-5 criteria for any dependence syndrome) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
* History of IV drug use.
* Current recreational use of ketamine.
* A positive urine drug screen on or after the screening visit during their active involvement in the study for ketamine, opiates, methadone, cocaine, amphetamines, benzodiazepines or cannabinoids.
* History of nonresponse or intolerance to ketamine.
* Significant uncontrolled physical illness particularly if it may affect the brain or glutamatergic system (blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure or severe chronic obstructive lung disease, autonomic neuropathies and active malignancy).
* Significant history of cardiovascular or cerebrovascular illness which may compromise the safety of ketamine use (myocardial infarction, heart failure, valvulopathy, stroke or transient ischaemic attack). Subjects with allergies and sensitivities to ketamine or similar compounds will also be excluded.
* Inability to provide a screening blood sample, urine sample or electrocardiogram.
* Biochemical abnormalities (defined as falling outside the normal reference range) as evaluated by a full blood count, and full biochemistry profile. Biochemical abnormalities must also be determined as clinically significant by a medical doctor to fulfil the criterion for exclusion.
* Electrocardiographic abnormalities, defined as any abnormality that is not normal sinus rhythm and determined as clinically significant by a medical doctor.
* Women of childbearing potential not using adequate contraception.
* Pregnant or breast-feeding women.
* Any previous neurosurgery or neurological disorder, including epilepsy
* History of head injury resulting in unconsciousness lasting at least 1 hour
* Any contraindications for MRI
* Use of compounds that may be affected by the use of ketamine (diazepam, warfarin, carbamazepine, phenytoin, theophylline and levothyroxine).
* Unwilling or unable to comply with the Lifestyle guidelines.

The following will be reasons for exclusion from analysis:

* Excessive head motion on resting state scan (Framewise displacement of 0.5mm on >20% of scans)
* Images not passing quality control as set out in the analysis plan
* Any side effects during the scan which could potentially impact interpretability of findings (e.g. nausea)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Glutamate | Changes will be in the same session comparing the ketamine infusion period to the pre-ketamine infusion baseline
  Compare changes in glutamate and GLX (glutamate +glutamine), referenced to total creatine (tCr), during ketamine infusion as measured by functional magnetic resonance spectroscopy (1H-fMRS) for naltrexone versus placebo pre-treatment conditions.
  Hypothesis: There will be a significant increase in glutamate measures during ketamine administration compared to a resting baseline condition in a medial prefrontal cortex (mPFC) /anterior cingulate cortex (ACC) region. Pre-treatment with naltrexone will attenuate this increase.

SECONDARY OUTCOMES:
Change in Resting State Functional Connectivity | Changes will be in the same session comparing post-infusion (immediately after ketamine infusion) to the pre-ketamine infusion baseline
  Compare changes in functional connectivity as measured by resting state-fMRI post-ketamine administration for naltrexone versus placebo pre-treatment conditions.
  Hypotheses:
  1. Ketamine administration will lead to significant reductions in functional brain connectivity between the subgenual anterior cingulate cortex (sgACC), default mode network (DMN) regions of interest (mPFC and posterior cingulate cortex (PCC)), thalamus, insula and ventral tegmental area (VTA) compared to a resting baseline condition. Pre-treatment with naltrexone will attenuate these reductions.
  2. Ketamine administration will lead to a significant increase in functional brain connectivity between the sgACC and dorsolateral prefrontal cortex (DLPFC) compared to a resting baseline condition. Pre-treatment with naltrexone will attenuate this increase.
Change in Cerebral Blood Flow | Changes will be in the same session comparing data collected 30 minutes after the ketamine infusion commences to the pre-ketamine infusion baseline
  Compare changes in cerebral blood flow during ketamine infusion as measured by arterial spin labelling (ASL) for naltrexone versus placebo pre-treatment conditions.
  Hypothesis: Ketamine administration will lead to a significant increase in CBF in sgACC, pregenual ACC (pgACC), dorsal ACC (dACC) and thalamus regions of interest compared to a resting baseline condition. Pre-treatment with naltrexone will attenuate these increases.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jelen LA, Lythgoe DJ, Stone JM, Young AH, Mehta MA. Effect of naltrexone pretreatment on ketamine-induced glutamatergic activity and symptoms of depression: a randomized crossover study. Nat Med. 2025 Sep;31(9):2958-2966. doi: 10.1038/s41591-025-03800-w. Epub 2025 Jul 24. PMID 40707608